CLINICAL TRIAL: NCT02279173
Title: A Single Arm, Open-label, Long-term Efficacy and Safety Study of Romiplostim in Thrombocytopenic Pediatric Subjects With Immune Thrombocytopenia (ITP)
Brief Title: Long-term Study of Romiplostim in Thrombocytopenic Pediatric Patients With Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101221; 2011-005019-96 (EudraCT Number)
Record Dates: First submitted 2014-10-01; First posted 2014-10-30 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Immune Thrombocytopenia
Keywords: Pediatric; Immune Thrombocytopenia; Amgen
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romiplostim (Experimental): Participants received romiplostim administered weekly by subcutaneous injection for up to 3 years. The starting dose was 1 µg/kg titrated in 1 µg/kg increments up to a maximum of 10 µg/kg to reach a target platelet count ≥ 50 x 10⁹/L.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Romiplostim subcutaneous weekly injection
  Other Names: Nplate

SUMMARY:
This is a phase 3b single arm, open label, multicenter study describing the percentage of time pediatric participants with ITP have a platelet response while receiving romiplostim, defined as a platelet count ≥ 50 x 10^9/L in the absence of ITP rescue medications for the past 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary ITP according to The American Society of Hematology (ASH) Guidelines at least 6 months before screening, regardless of splenectomy status
* Age ≥ 1 year and < 18 years of age
* Refractory to prior ITP therapy, relapsed after at prior ITP therapy, or be ineligible for other therapies. Examples of prior therapy include: corticosteroids, intravenous Immunoglobulin (IVIG), anti-D immunoglobulin, platelet transfusions.
* Platelet count ≤ 30 x10^9/L or is experiencing uncontrolled bleeding
* Has provided informed consent before any study-specific procedure;
* Adequate hematologic, renal, and liver function during screening:

  * Hemoglobin > 10.0 g/dL
  * Serum creatinine ≤ 1.5 x the upper limit of normal (ULN)
  * Total serum bilirubin ≤ 1.5 x the ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x the ULN
* For the EU, Switzerland and Turkey protocol supplement, subject must agree to a scheduled bone marrow biopsy and aspirate at Year 1 or Year 2 following romiplostim treatment and any unscheduled biopsies if clinically indicated
* For the EU, Switzerland and Turkey protocol supplement, a reticulin grade of 0, 1, 2, or 3 according to the modified Bauermeister grading scale, as assessed by central laboratory from a bone marrow biopsy performed within 1 year prior to planned first dose of romiplostim or consent to a pre-treatment bone marrow biopsy and aspirate prior to planned first dose of romiplostim

Exclusion Criteria:

* History of a bone marrow stem cell disorder (Any abnormal bone marrow findings other than those typical of ITP must be approved by Amgen before a subject may be enrolled)
* Prior bone marrow transplant or peripheral blood progenitor cell transplant
* Active or prior malignancy except non-melanoma skin cancers within the last 5 years
* History of myelodysplastic syndrome
* History of bleeding diathesis
* History of congenital thrombocytopenia
* History of Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV)
* History of systemic lupus erythematosus, Evans syndrome, or autoimmune neutropenia
* History of antiphospholipid antibody syndrome or known positive for lupus anticoagulant
* History of disseminated intravascular coagulation, hemolytic uremic syndrome, or thrombotic thrombocytopenic purpura
* History of venous thromboembolism or thrombotic events
* Previous use of romiplostim or previous use of eltrombopag within 4 weeks of enrollment
* Previous use of pegylated recombinant human megakaryocyte growth and development factor (PEG-rHuMGDF), recombinant human thrombopoietin (rHuTPO) or any other platelet producing agent
* Rituximab (for any indication) or 6-mercaptopurine within 8 weeks of enrollment, or anticipated use at any time during the study
* Splenectomy within 4 weeks of the screening visit
* Alkylating agents within 8 weeks before the screening visit or anticipated use during the time of the proposed study
* Vaccinations known to decrease platelet counts within 8 weeks before the screening visit
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending investigational study
* Will have investigational procedures while enrolled on study
* Female subject of child bearing potential (defined as having first menses) not willing to use, in combination with her partner highly effective methods of birth control during treatment and for 1 month after the end of treatment
* Subject is pregnant or breast feeding, or might become pregnant within 1 month after the end of treatment
* Subject has known hypersensitivity to any recombinant Escherichia coli derived product (eg, Infergen®, Neupogen®, somatropin, and Actimmune®)
* Has previously enrolled into this study
* Will not be available for protocol-required study visits or procedures, to the best of the subject's and investigator's knowledge
* Any kind of disorder that, may compromise the subject to give written informed consent and/or to comply with all required study procedures

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 203 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (73):
- United States (16):
  - Research Site, Roseville, California
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Randwick, New South Wales
  - Research Site, South Brisbane, Queensland
  - Research Site, Parkville, Victoria
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (3):
  - Research Site, Belém, Pará
  - Research Site, Jaú, São Paulo
  - Research Site, São Paulo, São Paulo
- Canada (3):
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Olomouc
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
- France (4):
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Vandœuvre-lès-Nancy
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
- Israel (6):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petach Tikvah
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Research Site, Monterrey, Nuevo León, Mexico
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Zabrze
- Russia (5):
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Volgograd
- South Africa (4):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Parktown, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Tygerberg, Western Cape
- Spain (4):
  - Research Site, Barcelona, Catalonia
  - Research Site, Esplugues de Llobregat, Catalonia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Turkey (Türkiye) (3):
  - Research Site, Adana
  - Research Site, Antalya
  - Research Site, Izmir
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Tarantino MD, Despotovic J, Roy J, Grainger J, Cooper N, Beam D, Raj A, Maschan A, Kim J, Eisen M. Romiplostim treatment for children with immune thrombocytopenia: Results of an integrated database of five clinical trials. Pediatr Blood Cancer. 2020 Nov;67(11):e28630. doi: 10.1002/pbc.28630. Epub 2020 Sep 9. PMID 32902132
- [Background] Grainger J, Bussel J, Tarantino M, Cooper N, Beam D, Despotovic J, Maschan A, Wang K, Eisen M, Bowers C. A single-arm, long-term efficacy and safety study of subcutaneous romiplostim in children with immune thrombocytopenia. Blood Adv. 2023 Feb 14;7(3):396-405. doi: 10.1182/bloodadvances.2021006014. PMID 35413092
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with immune thrombocytopenic purpura (ITP) and platelet counts ≤ 30×10⁹/L or uncontrolled bleeding were enrolled from December 2014 to August 2016 at 66 centers in 16 countries worldwide, including Eastern Europe (44%), Western Europe (25%), and US/Canada (21%).
Pre-assignment Details: All participants were assigned to receive weekly romiplostim.
  A subset of participants enrolled under a protocol supplement in the European Union (EU), Switzerland, and Turkey were enrolled into the following 2 cohorts:
  * bone marrow biopsy and aspirate at baseline and year 1
  * bone marrow biopsy and aspirate at baseline and year 2
Period: Overall Study
Arm/Group | Romiplostim
Started | 203
Received Treatment | 203
Enrolled Under Protocol Supplement | 79
Completed | 109
Not Completed | 94
Not completed — Protocol-specified Criteria | 67
Not completed — Withdrawal by Subject | 20
Not completed — Decision by Sponsor | 4
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 203
Age, Continuous [Median (Full Range); unit: years] | 10.0 [1 to 17]
Age, Customized [Count of Participants; unit: Participants]
  ≥ 1 to < 6 years | 49
  ≥ 6 to < 12 years | 81
  ≥ 12 to < 18 years | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 12
  Black or African American | 11
  Multiple | 1
  Native Hawaiian or Other Pacific Islander | 0
  Other, Not Specified | 11
  White | 164
Years Since ITP Diagnosis [Median (Full Range); unit: years] — Population: Participants with available data
  years | 1.75 [0.5 to 13.8]
Age at ITP Diagnosis [Median (Full Range); unit: years] — Population: Participants with available data
  years | 5.97 [0.6 to 17.3]
Splenectomy Done [Count of Participants; unit: Participants]
  Yes | 10
  No | 193
Platelet Count [Median (Full Range); unit: 10⁹ cells/L] — Population: Participants with available data
  10⁹ cells/L | 14.00 [1.5 to 265.0]
Number of Prior ITP Treatments [Median (Full Range); unit: prior ITP treatments] — Population: Participants with available data
  prior ITP treatments | 2.0 [1 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time With a Platelet Response During the First 6 Months of Treatment
Description: Platelet response was defined as a platelet count of ≥ 50 x 10⁹/L with no rescue medication use for ITP in the past 4 weeks.
  Monthly platelet response was calculated based on the median platelet count during each month. For each participant, the percentage of time with platelet response during the first 6 months was calculated as the number of months a platelet response was observed divided by the total number of months response was assessed.
Time Frame: Week 2 to Month 6, platelet response was assessed every week.
Population: The efficacy analysis set included all enrolled participants who received at least 1 dose of romiplostim
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Romiplostim
Number analyzed (Participants) | 203
percentage of time | 50.00 [16.67 to 83.33]

2. Primary Outcome: Percentage of Participants Who Developed Collagen After Exposure to Romiplostim
Description: The percentage of participants who developed collagen as evidenced by trichrome staining, defined as a Grade 4 on the modified Bauermeister grading scale:
  Grade 0: No reticulin fibers demonstrable
  Grade 1: Occasional fine individual fibers and foci of a fine fiber network
  Grade 2: Fine fiber network throughout most of the section; no coarse fibers
  Grade 3: Diffuse fiber network with scattered thick coarse fibers but no mature collagen (negative to trichrome staining)
  Grade 4: Diffuse, often course fiber network with areas of collagenization (positive trichrome staining)
Time Frame: Year 1 (Cohort 1) and year 2 (Cohort 2)
Population: The bone marrow analysis set includes participants who received at least 1 dose of romiplostim, who were recruited within the protocol supplement for the EU, Switzerland and Turkey and who had at least 1 bone marrow biopsy during the study after initiation of study treatment. Participants with available core biopsy results are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1: Participants enrolled under the protocol supplement in the EU, Switzerland, or Turkey received weekly romiplostim for 3 years and had a bone marrow biopsy at baseline and year 1.
- Cohort 2: Participants enrolled under the protocol supplement in the EU, Switzerland, or Turkey received weekly romiplostim for 3 years and had a bone marrow biopsy at baseline and year 2.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 36
percentage of participants | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 9.7]

3. Secondary Outcome: Percentage of Time With a Platelet Response During the Overall Treatment Period
Description: Platelet response was defined as a platelet count of ≥ 50 x 10⁹/L with no rescue medication use in the past 4 weeks.
  Monthly platelet response was calculated based on the median platelet count during each month. For each participant, the percentage of time with platelet response was calculated as the number of months a platelet response was observed divided by the total number of months response was assessed.
Time Frame: From week 2 to the end of the treatment period, 36 months
Population: Efficacy analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Romiplostim
Number analyzed (Participants) | 203
percentage of time | 78.21 [26.67 to 90.39]

4. Secondary Outcome: Percentage of Time With an Increase in Platelet Count ≥ 20 x 10⁹ Cells/L Above Baseline
Description: The percentage of time with an increase in platelet count ≥ 20 x 10⁹ cells/L above baseline from week 2 until the end of the treatment period without rescue medication use within the past 4 weeks.
  For each participant, the percentage of time with an increase in platelet count ≥ 20 x10⁹ cells/L above baseline was calculated as the number of months the median platelet count was ≥ 20 x10⁹ cells/L above baseline divided by the total number of months assessed.
Time Frame: Baseline and from week 2 to month 36
Population: Efficacy analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Romiplostim
Number analyzed (Participants) | 203
percentage of time | 80.13 [39.13 to 92.31]

5. Secondary Outcome: Number of Participants Reporting Use of Rescue Medications for ITP During the Treatment Period
Description: Rescue medication is defined as any medication or transfusion, other than romiplostim and excluded medications, that is administered after enrollment to the participant with the intent of raising platelet counts or to prevent bleeding and includes concomitant medications for ITP in which the dose and/or schedule was increased. Permitted rescue medications included the following:
  * corticosteroids
  * platelet transfusions
  * Intravenous immunoglobulin (IVIG)
  * azathioprine
  * anti-D immunoglobulin
  * danazol
Time Frame: From first dose of romiplostim to the end of the treatment period, 36 months
Population: Efficacy analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 203
Participants | 60

6. Secondary Outcome: Number of Participants Who Developed Anti-Romiplostim or Anti-Thrombopoietin Neutralizing Antibodies
Description: Blood samples were first tested for the presence of binding antibodies to romiplostim or the peptide portion of romiplostim, and to endogenous thrombopoietin (eTPO). Samples testing positive for binding antibodies were then tested for neutralizing antibodies by assessing their ability to neutralize romiplostim and/or eTPO in a cell-based bioassay.
  Participants who developed neutralizing antibodies are those who had a postbaseline positive result with a negative or no result at baseline. Transient is defined as a negative result at the participant's last time point tested within the study period.
Time Frame: Week 12, week 52 and every 24 weeks thereafter up to month 36
Population: Participants who received at least 1 dose of romiplostim and with a post-baseline antibody result.
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 203
Participants
  Anti-romiplostim neutralizing antibodies | 7
  Transient anti-romiplostim neutralizing antibodies | 4
  Anti-eTPO neutralizing antibodies | 1
  Transient anti-eTPO neutralizing antibodies | 1

7. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participant, which does not necessarily have a causal relationship with study treatment.
  A serious adverse event (SAE) was defined as an AE that met at least 1 of the following criteria:
  * fatal
  * life threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event Adverse events were graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 grading scale, where Grade 1 = mild AE; Grade 2 = moderate AE; Grade 3 = severe AE; Grade 4 = life-threatening or disabling; Grade 5 = death related to AE.
Time Frame: SAEs were collected from Screening through end-of-study follow-up (up to 38 months). Nonserious AEs were collected from first to last dose of study drug during the treatment period (up to 36 months).
Population: Participants who received at least 1 dose of romiplostim
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 203
Participants
  Any adverse event (AE) | 193
  Serious adverse events (SAE) | 60
  AEs leading to discontinuation of romiplostim | 15
  Adverse event Grade ≥ 3 | 66
  Adverse event Grade ≥ 4 | 19
  Adverse event Grade ≥ 5 | 0
  Treatment-related adverse events (TRAE) | 56
  Treatment-related serious adverse events | 8
  TRAEs leading to discontinuation of romiplostim | 8
  Treatment-related adverse events Grade ≥ 3 | 8
  Treatment-related adverse events Grade ≥ 4 | 0
  Treatment-related adverse events Grade ≥ 5 | 0

8. Primary Outcome: Percentage of Participants With Increased Modified Bauermeister Grade
Description: The percentage of participants with an increased modified Bauermeister grade defined as an increase by ≥ 2 severity grades or an increase to grade 4 (i.e., grade 0 to 2-4, grade 1 to 3-4, grade 2 to 4, or grade 3 to 4 over baseline). The modified Bauermeister grading scale:
  Grade 0: No reticulin fibers demonstrable
  Grade 1: Occasional fine individual fibers and foci of a fine fiber network
  Grade 2: Fine fiber network throughout most of the section; no coarse fibers
  Grade 3: Diffuse fiber network with scattered thick coarse fibers but no mature collagen (negative to trichrome staining)
  Grade 4: Diffuse, often course fiber network with areas of collagenization (positive trichrome staining)
  Participants without an evaluable baseline result were assumed to have a baseline modified Bauermeister score of 0.
Time Frame: Baseline, year 1 (Cohort 1) and year 2 (Cohort 2)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 36
percentage of participants | 3.7 [0.1 to 19.0] | 0.0 [0.0 to 9.7]

9. Primary Outcome: Percentage of Participants Who Developed Bone Marrow Abnormalities
Description: The percentage of participants with bone marrow abnormalities (eg, myelodysplastic syndrome, monosomy 7) based on analysis of bone marrow biopsy and aspirate samples using cytogenetics and fluorescence in situ hybridization.
Time Frame: Year 1 (Cohort 1) and year 2 (Cohort 2)
Population: Bone marrow analysis set participants with an on-study bone marrow abnormality assessment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 31
percentage of participants | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 11.2]

10. Secondary Outcome: Percentage of Participants Who Developed Increased Reticulin
Description: The percentage of participants with increased reticulin as evidenced by silver staining and defined as any increase from baseline in the modified Bauermeister grade:
  Grade 0: No reticulin fibers demonstrable
  Grade 1: Occasional fine individual fibers and foci of a fine fiber network
  Grade 2: Fine fiber network throughout most of the section; no coarse fibers
  Grade 3: Diffuse fiber network with scattered thick coarse fibers but no mature collagen (negative to trichrome staining)
  Grade 4: Diffuse, often course fiber network with areas of collagenization (positive trichrome staining)
  Participants without an evaluable baseline result were assumed to have a baseline modified Bauermeister score of 0.
Time Frame: Baseline, year 1 (Cohort 1) and year 2 (Cohort 2)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 36
percentage of participants | 18.5 [6.3 to 38.1] | 47.2 [30.4 to 64.5]

ADVERSE EVENTS:
Time Frame: SAEs were collected from Screening through end-of-study follow-up (up to 38 months). Nonserious AEs were collected from first to last dose of study drug during the treatment period (up to 36 months).
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Romiplostim
All-Cause Mortality (participants affected / at risk) | 0/203
Serious Adverse Events (participants affected / at risk) | 60/203
Other Adverse Events (participants affected / at risk) | 183/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=203)
Anaemia (Blood and lymphatic system disorders) | 2
Evans syndrome (Blood and lymphatic system disorders) | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 3
Lymphadenitis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Gastroenteritis rotavirus (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Otitis externa (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Staphylococcal abscess (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Arthroscopy (Investigations) | 1
Blood urine present (Investigations) | 1
Neutralising antibodies positive (Investigations) | 4
Platelet count decreased (Investigations) | 10
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Lupus nephritis (Renal and urinary disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Polymenorrhoea (Reproductive system and breast disorders) | 1
Varicocele (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=203)
Anaemia (Blood and lymphatic system disorders) | 13
Ear pain (Ear and labyrinth disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 29
Abdominal pain upper (Gastrointestinal disorders) | 39
Diarrhoea (Gastrointestinal disorders) | 38
Gingival bleeding (Gastrointestinal disorders) | 21
Mouth haemorrhage (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 37
Vomiting (Gastrointestinal disorders) | 47
Fatigue (General disorders) | 19
Pyrexia (General disorders) | 65
Hypersensitivity (Immune system disorders) | 12
Conjunctivitis (Infections and infestations) | 13
Ear infection (Infections and infestations) | 15
Gastroenteritis (Infections and infestations) | 19
Influenza (Infections and infestations) | 18
Nasopharyngitis (Infections and infestations) | 75
Pharyngitis (Infections and infestations) | 32
Rhinitis (Infections and infestations) | 40
Tonsillitis (Infections and infestations) | 15
Upper respiratory tract infection (Infections and infestations) | 39
Viral infection (Infections and infestations) | 21
Contusion (Injury, poisoning and procedural complications) | 40
Fall (Injury, poisoning and procedural complications) | 13
Skin laceration (Injury, poisoning and procedural complications) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 78
Cough (Respiratory, thoracic and mediastinal disorders) | 52
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 77
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 37
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 27
Ecchymosis (Skin and subcutaneous tissue disorders) | 19
Petechiae (Skin and subcutaneous tissue disorders) | 48
Rash (Skin and subcutaneous tissue disorders) | 27
Haematoma (Vascular disorders) | 42
Sinusitis (Infections and infestations) | 11
Limb injury (Injury, poisoning and procedural complications) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT02279173/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT02279173/SAP_001.pdf